CLINICAL TRIAL: NCT01833871
Title: Uterine Artery Doppler and Three Dimensional Power Doppler in the Diagnosis of Myometrial Masses
Brief Title: The Use of Doppler to Diagnose Myometrial Masses
Acronym: 3D
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Elkattan, Dr., Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Protocol200
Record Dates: First submitted 2013-04-04; First posted 2013-04-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Uterine Masses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- myometrial fibroid/adenomyoma (Experimental): Patients scheduled for myomectomy or hysterectomy with preoperative diagnosis of uterine myoma, adenomyosis or both by ultrasound .Trans-vaginal 3D power Doppler and uterine artery doppler will be done for all participants prior to surgery.
  Interventions: Other: Three dimensional Power Doppler to the myometrial mass; Other: Uterine artery Doppler

INTERVENTIONS:
Other: Three dimensional Power Doppler to the myometrial mass — Trans-vaginal 3D power Doppler Ultrasonographic examination will be done for all participants prior to surgery. The ultrasonographic examination will provide data related to lesion size, lesion volume, vascular location (location), vascular index (VI), flow index (FI), and vascular-flow index (VFI). The region of interest will include the entire region of the uterine mass. The virtual organ computer aided analysis (VOCAL) software for the analysis of 3D power Doppler histograms will be used with computer algorithms to form indices of blood flow and vascularization. All data will be collected and compared with the post operative histopathology results.
Other: Uterine artery Doppler — uterine artery Doppler indices(RI,PI) are measured for all cases with myometrial mass

SUMMARY:
Colour Doppler sonography has also been evaluated in differentiating adenomyosis from fibroids. Two dimensional color Doppler ultrasound revealed that 87% of adenomyosis cases had vessel distributions different from those found in leiomyoma cases, in addition to a high pulsatility index (PI) .Adenomyotic lesions had randomly scattered vessels or intratumoral signals while leiomyomas usually had peripheral scattered or outer feeding vessels.

DETAILED DESCRIPTION:
Because it is more sensitive, less angle-dependent, and not susceptible to aliasing , power Doppler Sonography has the potential to detect fluctuations in blood flow , with results superior to those of frequency-based color Doppler sonography, particularly in situations of low-velocity blood flow. Three dimensional power Doppler ultrasonography can be applied to differentiate between uterine adenomyosis and leiomyoma ,and it may reduce the number of false positives by detailed investigations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 & 60 years.
* Asymptomatic pts which discover the mass accidentally .
* Patients with symptoms like menorrhagia, menometrorrhagia, dysmenorrheal , abdominal masses.
* Patients scheduled for hysterectomy(abdominal/vaginal or Laparoscopic)
* Patients scheduled for myomectomy.

Exclusion Criteria:

* Pregnant patients
* Age over 60 or under 20years.
* Conservative management (Non surgical)

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Power Doppler Vascular indices | 9 months
  The ultrasonographic examination will provide data related to lesion size, lesion volume, uterine artery doppler indices and vascular location (location), vascular index (VI), flow index (FI), and vascular-flow index (VFI). The region of interest will include the entire region of the uterine mass. The virtual organ computer aided analysis (VOCAL) software for the analysis of 3D power Doppler histograms will be used with computer algorithms to form indices of blood flow and vascularization. All data will be collected and compared with the post operative histopathology results.
Uterine artery doppler indices in fibroids in relation to adenomyosis | 9 months
  Uterine artery doppler indices(RI,PI) in fibroids in relation to adenomyosis

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt